CLINICAL TRIAL: NCT01950663
Title: RETeval Calibration / Validation Study - Diabetic Retinopathy
Brief Title: RETeval Study for Diabetic Retinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inoveon Corporation (Industry)
Collaborators: LKC Technologies, Inc. (Industry); National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Stephen R Fransen, MD, Chief Medical Officer, Inoveon Corporation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3032; R44EY021121 (NIH)
Record Dates: First submitted 2013-09-05; First posted 2013-09-25 (Estimated); Results first posted 2017-05-09 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-05

CONDITIONS: Diabetic Retinopathy
Keywords: Diagnostic Equipment; Validation Studies
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RETeval (Experimental): RETeval is a new handheld device intended to detect vision threatening diabetic retinopathy by measuring the response of the retina to a flash of light.
  Interventions: Device: RETeval

INTERVENTIONS:
Device: RETeval — RETeval is a new handheld device intended to detect vision threatening diabetic retinopathy by measuring the response of the retina to a flash of light.

SUMMARY:
RETeval is a new handheld device intended to detect vision threatening diabetic retinopathy. The purpose of this study is to calibrate RETeval, and then measure its ability to detect vision threatening diabetic retinopathy. Early Treatment Diabetic Retinopathy Study (ETDRS) 7-field, dilated, stereo, color fundus photography, read according to the ETDRS protocol, will be used as the gold standard.

DETAILED DESCRIPTION:
Diabetic retinopathy is the leading cause of preventable blindness in working age Americans. The associated loss of quality of life, and the economic loss from health care costs and lost productivity, are staggering. This burden is increasing rapidly as the epidemic of diabetes continues. In the developing world, diabetic retinopathy is expected to become the leading cause of preventable blindness since the prevalence of diabetes correlates closely with the dietary changes, obesity, and sedentary lifestyles that accompany economic development.

Half of all people with proliferative diabetic retinopathy will be blind within five years. With proven laser and intravitreal drug therapy this risk is reduced to less than 5%, a ten-fold decrease in risk. One third of all people with diabetic macular edema will suffer moderate visual loss in three years. With proven therapy this risk is reduced to less than 10%, a three-fold decrease in risk. Nonetheless, diabetic retinopathy remains the leading cause of preventable blindness in working age Americans.

Excellent diabetes control prevents or significantly reduces the development and progression of diabetic retinopathy but this approach requires difficult lifestyle changes. Therefore, timely identification of patients at risk for blindness, and assuring they receive proven care, are essential to eliminate blindness from diabetic retinopathy. Unfortunately, despite decades of public health awareness campaigns and programs, only 56.9% of US patients with diabetes received universally recommended eye evaluations in 2011.

One reason for this failure is the complexity of existing methods for diabetic retinopathy testing. To be effective, accurate testing should be available in the primary care physician's office since the need for an additional visit to an ophthalmologist is another reason universal testing has failed. To succeed in the primary care physician's office, existing personnel, with minimal training, must be able to accurately and easily test patients. The testing method must take little time and require no additional space since efficient time and space utilization are critical in primary care settings. It must meet quality measures used by Medicare and other payors to award financial incentives. Finally, it must be reimbursed at a favorable level.

RETeval is LKC Technologies' new, handheld, non-invasive, device that measures full-field electroretinogram (ERG) cone b-wave photopic flicker implicit times quickly and easily in a primary care setting. RETeval is simple to use and takes less than five minutes for most patients. It is a handheld device that requires no additional space. Based on published literature, the implicit time is significantly delayed in eyes with severe non proliferative diabetic retinopathy (NPDR) and proliferative diabetic retinopathy (PDR) relative to eyes with milder forms of DR. These findings suggest that the photopic ERG implicit time can be a good indicator for the objective evaluation of the severity of DR ranging from mild NPDR to PDR.

This study will measure the accuracy of the RETeval device. ETDRS 7-field, dilated, stereo, color fundus photography, read according to the ETDRS protocol, will be used as the gold standard. Cone b-wave photopic flicker implicit time, measured by the RETeval device, and ETDRS photography, will be performed during a single visit. A random sample of the results, the calibration set, will be used to calibrate the referral threshold for the RETeval device. The remaining results, the validation set, will be used as an independent validation to assess accuracy. If RETeval is accurate, and is accepted as a quality measure meeting performance standards, it will be an ideal method to test for retinopathy in patients with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with diabetes and treated with at least one oral hypoglycemic medication or insulin
* Eighteen years or older

Exclusion Criteria:

* History of photosensitive epilepsy
* Previous laser or drug treatment for diabetic retinopathy or macular edema
* Eye diseases other than diabetic retinopathy or macular edema that, in the opinion of the recruiting ophthalmologist, may affect the electroretinogram or result in ungradable Early Treatment Diabetic Retinopathy Study Protocol images.
* Inability or unwillingness of the subject or legal guardian/representative to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Actual)
Dates: Start 2013-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen R Fransen, MD, Principal Investigator — Inoveon Corporation
Locations (2):
- United States (2):
  - Atlanta VA Medical Center, Decatur, Georgia
  - Oklahoma City VA Medical Center, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RETeval
Started | 468
Completed | 467
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | RETeval
Number analyzed (Participants) | 467
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 409
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 458
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 24
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 184
  White | 243
  More than one race | 0
  Unknown or Not Reported | 14
Region of Enrollment [Number; unit: participants]
  United States | 467

OUTCOME MEASURES:

1. Primary Outcome: Per Patient Referral Accuracy
Description: Accuracy will be reported as count of participants with referral status correctly identified, sensitivity, and specificity, with ETDRS photography and reading as the gold standard.
Time Frame: During a single visit, implicit time, measured by the RETeval device, and ETDRS photography, will be performed to support the analysis of the accuracy of the RETeval device.
Population: Participants with gradeable fundus photos and RETeval measurements
Measure: Count of Participants; unit: Participants
Arm/Group | RETeval
Number analyzed (Participants) | 401
Participants | 318

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | RETeval
All-Cause Mortality (participants affected / at risk) | 0/468
Serious Adverse Events (participants affected / at risk) | 0/468
Other Adverse Events (participants affected / at risk) | 0/468

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No